CLINICAL TRIAL: NCT00990639
Title: Beneficial Effect of Angiotensin-blocking Agent Candesartan on Alcoholic Liver Fibrosis: A Randomized Controlled Trial
Brief Title: Effect of Candesartan in Alcoholic Liver Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Soon Koo Baik/ Yonsei University Wonju College of Medicine Department of Internal Medicine Devision of Gastroenterology and Hepatology, Yonsei University Wonju College of Medicine Department of Internal Medicine Devision of Gastroenterology and Hepatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YWhep091
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Alcoholic Liver Disease
Keywords: hepatic fibrosis; angiotensin II blocking agents; alcoholic liver disease
MeSH Terms: conditions — Liver Diseases, Alcoholic; Liver Cirrhosis | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- candesartan+UDCA group (Experimental): oral candesartan(8 mg/day) in addition to ursodeoxycholic acid (UDCA, 600 mg/day) for 6 months
  Interventions: Drug: candesartan for hepatic fibrosis
- UDCA group (Placebo Comparator): ursodeoxycholic acid(UDCA,600 mg/day)only for 6 months
  Interventions: Drug: candesartan for hepatic fibrosis

INTERVENTIONS:
Drug: candesartan for hepatic fibrosis — Candesartan group(42 patients): oral candesartan at a daily dose of 8 mgin addition to ursodeoxycholic acid (UDCA, 600 mg/day) for 6 months.
  UDCA group(43 patients): oral ursodeoxycholic acid (UDCA, 600 mg/day) only for 6 months
  Other Names: atacand for hepatic fibrosis

SUMMARY:
Background:

Alcohol is one of principal causes of hepatic fibrosis. Although the most effective treatment for alcoholic hepatic fibrosis is abstinence of alcohol consumption, additive treatment to reduce the accumulation of scar tissue can accelerate the improvement of hepatic fibrosis in alcoholic liver disease. The renin-angiotensin system can be an attractive antifibrotic target in liver. Several lines of evidence indicate that overproduction of angiotensin II(ANG II) in chronic liver injury stimulates the activation of hepatic stellate cells(HSCs) attributed to fibrogenesis. Additionally, the antifibrotic effect of ANG II blocking agent has been shown in various animal models and hepatitis C patients. Hence, drugs that inhibit the renin-angiotensin system have promise in ameliorating hepatic fibrosis in chronic liver injury. However, no study has been conducted in patients with alcoholic liver disease to evaluate the effect ANG II type I receptor blocking agent on hepatic fibrosis.

Aim:

This study aimed to investigate the safety and the efficacy of chronic administration of candesartan to hepatic fibrosis patients with alcoholic liver disease.

Methods

1) Patients with liver fibrosis(F2) were randomized to receive either the angiotensin receptor blocker(ARB), candesartan(8 mg/day) with ursodeoxycholic acid(UDCA)(600 mg/day)(n = 42), or UDCA alone(n = 43) as control for 6 months. 2)All enrolled patients underwent liver biopsies twice for measurement of fibrosis score, area of fibrosis and alpha-smooth muscle actin(SMA) positive and hydroxyproline. 3) Transforming growth factor-beta1(TGF-beta1), collagen-1, angiotensin II type I receptor(AT1-R), tissue inhibitor of metalloproteinase-1(TIMP-1), Rac1 and p22phox which represent oxidant stress were also measured by real-time RT-PCR before and after 6 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of alcoholic liver disease
* METAVIR fibrosis score ≥ 2 in liver biopsy
* Alcohol intake has stop during at least 6 months until study enrollment

Exclusion Criteria:

* Hepatocellular carcinoma or other malignancy
* Clinically decompensated cirrhosis (Total bilirubin ≥ 5mg/dL or variceal hemorrhage or ascites development or hepatic encephalopathy developement)
* Chronic liver disease related with other causes except alcohol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improvement of histologic grade of hepatic fibrosis | 6 month later

SECONDARY OUTCOMES:
estimation of safety of candesartan in hepatic fibrosis | 6 month later

CONTACTS AND LOCATIONS:
Overall Officials: Soon Koo Baik, Professor, Principal Investigator — Yonsei University Wonju College of Medicine Department of Internal Medicine Devision of Gastroenterology and Hepatology
Locations (1):
- Yonsei University Wonju College of Medicine Wonju Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Background] Corey KE, Shah N, Misdraji J, Abu Dayyeh BK, Zheng H, Bhan AK, Chung RT. The effect of angiotensin-blocking agents on liver fibrosis in patients with hepatitis C. Liver Int. 2009 May;29(5):748-53. doi: 10.1111/j.1478-3231.2009.01973.x. Epub 2009 Feb 9. PMID 19220742
- [Background] Rimola A, Londono MC, Guevara G, Bruguera M, Navasa M, Forns X, Garcia-Retortillo M, Garcia-Valdecasas JC, Rodes J. Beneficial effect of angiotensin-blocking agents on graft fibrosis in hepatitis C recurrence after liver transplantation. Transplantation. 2004 Sep 15;78(5):686-91. doi: 10.1097/01.tp.0000128913.09774.ce. PMID 15371669
- [Background] Debernardi-Venon W, Martini S, Biasi F, Vizio B, Termine A, Poli G, Brunello F, Alessandria C, Bonardi R, Saracco G, Rizzetto M, Marzano A. AT1 receptor antagonist Candesartan in selected cirrhotic patients: effect on portal pressure and liver fibrosis markers. J Hepatol. 2007 Jun;46(6):1026-33. doi: 10.1016/j.jhep.2007.01.017. Epub 2007 Feb 9. PMID 17336417
- [Background] Terui Y, Saito T, Watanabe H, Togashi H, Kawata S, Kamada Y, Sakuta S. Effect of angiotensin receptor antagonist on liver fibrosis in early stages of chronic hepatitis C. Hepatology. 2002 Oct;36(4 Pt 1):1022. doi: 10.1053/jhep.2002.32679. No abstract available. PMID 12297856